CLINICAL TRIAL: NCT01451684
Title: Development of a Non-invasive Prenatal Test
Status: Completed | Type: Observational
Sponsor: Cindy Cisneros (Industry)
Responsible Party: Sponsor-Investigator, Cindy Cisneros, CRA, Roche Sequencing Solutions
Organization: Roche Sequencing Solutions (Industry)
Other Study IDs: TD003
Record Dates: First submitted 2011-10-10; First posted 2011-10-14 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Pregnancy
Keywords: pregnancy; fetus; euploid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study to aid in the development of a non-invasive prenatal test that may be used to aid in detection of fetal aneuploidy. Pregnant women will be recruited and asked to provide a blood sample to be used for general test development purposes.

DETAILED DESCRIPTION:
Blood samples and information collected for the study will be used for test development and quality control purposes. No test results will be communicated back to study subjects or their health care providers.

ELIGIBILITY:
Inclusion Criteria:

* Subject has singleton or twin pregnancy confirmed via evaluation by a healthcare provider
* Subject is able to provide informed consent
* Subject is ≥ 18 years of age
* Subject is at least 10 weeks gestation for general enrollment
* Subject has no known risk factors for chromosomal abnormalities of the fetus
* Subject has no suspected or confirmed fetal abnormalities

Exclusion Criteria:

* Subject is pregnant with more than two fetuses
* Subject is unwilling to undergo a blood draw

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include women who have a healthy pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2011-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Absence of chromosomal abnormality | At time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Roberts, Study Director — Ariosa Diagnostics
Locations (1):
- Ariosa Diagnostics, San Jose, California, United States